CLINICAL TRIAL: NCT07062705
Title: Comparative Effects of Neural Tissue Mobilization and Progressive Inhibition of Neuromuscular Structure (PINS) Technique on Pain, Range and Disability in Patients With Lumbar Radiculopathy.
Brief Title: Progressive Inhibition of Neuromuscular Structure and Neural Tissue Mobilization.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0168
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Lumbar Radiculopathy
Keywords: Pain; Range; Disability
MeSH Terms: conditions — Radiculopathy; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Inhibition of Neuromuscular Structure (Active Comparator): The index fingers of both hands were used to palpate two connected locations, referred to as main and endpoints. along a neuromuscular structure and were the most and least sensitive sections, respectively. After identifying the primary point-the area of greatest sensitivity-a moderate ischemic compression was also applied for 30 seconds using the index finger of the other hand. Next, a second sensitive point was located using the middle finger of the same hand, proximal to the endpoint, without releasing the pressure from the index finger. The index finger pressure was released and the middle finger pressure was kept constant without releasing the endpoint pressure when it was seen that the middle finger was more sensitive to pressure than the index finger.
  Interventions: Other: Progressive Inhibition of Neuromuscular Structure
- Neural Tissue Mobilization. (Active Comparator): The patient sat well back on the end of a plinth with thighs fully supported. The patient was asked to slump or sag while examiner maintains cervical spine in neutral position. Overpressure was applied to the lumbar and thoracic flexion in attempt to bow the spine rather than the hips. With spinal flexion position maintained, the patient was asked to bend his chin to chest and then overpressure in the same direction was added. The patient was asked to extend his knee actively. The patient was asked to dorsiflex his ankle.
  Interventions: Other: Neural Tissue Mobilization.

INTERVENTIONS:
Other: Progressive Inhibition of Neuromuscular Structure — The index fingers of both hands were used to palpate two connected locations, referred to as main and endpoints. The locations were located along a neuromuscular structure and were the most and least sensitive sections, respectively. Once an endpoint (region of least sensitivity) was identified, the index finger of one hand was used to provide a moderate ischemia compression; the pressure was kept constant until the course of therapy was finished. After identifying the primary point-the area of greatest sensitivity-a moderate ischemic compression was also applied for 30 seconds using the index finger of the other hand.
  Arms: Progressive Inhibition of Neuromuscular Structure
Other: Neural Tissue Mobilization. — The patient sat well back on the end of a plinth with thighs fully supported. The patient was asked to slump. Overpressure was applied to the lumbar and thoracic flexion in attempt to bow the spine rather than the hips. With spinal flexion position maintained, the patient was asked to bend his chin to chest and then overpressure in the same direction was added. The patient was asked to extend his knee actively. The patient was asked to dorsiflex his ankle. The therapist was maintaining the ankle dorsiflexion as a progression for technique. The number of these sequences was repeated several times,through which the amplitude of the technique was increased according to the patient response. The technique was progressed to a point where symptoms reproduced, or it was taken to a point where resistance of the movement was encountered.
  Arms: Neural Tissue Mobilization.

SUMMARY:
Lumbar radiculopathy is a neuromusculoskeletal condition that is characterized as radiating pain in the leg described as electric, burning, or sharp, and is associated with dermatomal or myotomal differences and tendon reflex abnormalities. Neural mobilization is a manual therapy technique designed to alleviate nerve pain and dysfunction by gently mobilizing the nerve along its pathway. The Progressive Inhibition of Neuromuscular Structures (PINS) technique is a therapeutic approach that aims to reduce pain and muscle tension by sequentially applying pressure to specific points along a muscle or nerve pathway. This study focuses on pain, range of motion and disability with these techniques in patients with lumbar radiculopathy.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial and will be conducted in Hassan healthcare centre Gujrat. Non-probability conveninet sampling technique will be used to collect the data. Sample size of 48 subjects (per group 16) with age group between 18-40 years will be taken. Individuals having radiculopathy at level of L5-S1 (unilateral radiculopathy) and pain in the distribution of sciatic nerve (leg-dominant symptoms). Outcome measure will be taken using Numeric pain rating scale (NPRS), Oswestry Disability Index (ODI), Sciatica Bothersomeness Index (SBI), Goniometer. An informed consent will be taken. Subjects will be selected on the basis of inclusion and exclusion criteria and will be equally divided into three groups. Both the Groups will receive Hot Pack, lumbar stabilization including curl ups and side bridging and stretching include hamstring stretch and piriformis stretch. Group A will receive PINS technique as per Dowling's guidelines. Group 2 will receive Neural mobilization technique. Groyup 3 will receive both PINS and neural mobilization technique. Outcome measures will be measured at baseline and after 4 weeks. Each group (both single and combined) will receive two treatments per week for 30 min each, for 4 weeks. Data analysis will be done by SPSS version 26.

ELIGIBILITY:
INCLUSION CRITERIA

* Age group between 18 and 40 years(.
* Both gender male and female.
* Participants diagnosed as having a chronic (lasting three months or longer) lumbar radiculopathy.
* Diagnosed patient of having radiculopathy at level of L4-L5 and L5-S1 lesion (unilateral radiculopathy).
* Radiating pain evoked by specific clinical tests, including slump and straight leg raise.

Exclusion Criteria:

* Individuals having bilateral lumbar radiculopathy.
* Spondylolysis/spondylolisthesis
* Mechanical systemic low back pain or neoplasmic and infectious processes.
* Participants with severe nerve root compression (non-ambulant/wheelchair-bound).
* Any sign or symptom of dementia or other cognitive impairments.
* Diagnosis of claudication, previous spinal surgery, pregnancy and presence of any of the spinal red flags.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-07-24 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
NUMERIC PAIN RATING SCALE (NPRS): | 4 weeks
  Low back and leg pain were measured using the numeric pain rating scale (NPRS), as has been used in various randomized controlled trials for NE and spinal pain. 41,42,48 The minimal detectable change for the NPRS is reported to be 2.1

SECONDARY OUTCOMES:
OSWESTRY DISABILITY INDEX (ODI): | 4 weeks
  The ODI assesses the impacts of low back pain or leg pain on the physical function and activities of daily living. It has been shown to have high levels of reliability, validity and responsiveness in patients with low back pain(20). A change of 5 points (10%) has been proposed as the minimal detectable change.

OTHER OUTCOMES:
Sciatica Bothersomeness Index (SBI): | 4 weeks
  This scale was used to assess the level of sciatica among participants. The scale's scores range from 0 to 24, with higher scores reflecting more severe sciatica bothersomeness. This scale has a high level of internal consistency reliability (Cronbach's alpha of 0.70) and test-retest reliability (ICC of 0.90); a change of 6.5 points is considered clinically significant

CONTACTS AND LOCATIONS:
Overall Officials: Muzna Munir, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Hassan Health Care Centre, Gujrat, Dhok Gujra, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olofson E, Gerona C, Estrada A, Duong J. Joint and Neural Mobilization for Pain Reduction in Radiculopathy Patients: Azusa Pacific University; 2023.
- [Background] Malik A, Ramsha M, Samad A. Outcomes of the butler neural mo-bilization technique and manual therapy for chronic low back pain in patients with lumbar radiculopathy: A cross-sectional comparative study. J Basic Clin Med Sci. 2022;1:3-11
- [Background] Divyasree S, Kumaresan A, Vishnuram S. Effect of Mckenzie lumbar extension exercise with TENS on lumbar radiculopathy. Biomedicine. 2023;43(3):1032-5.
- [Background] Danazumi MS, Ibrahim SU. Effectiveness of Progressive Inhibition of Neuromuscular Structures (PINS) and Spinal Mobilization with Leg Movement (SMWLM) in Lumbar Disk Herniation with Radiculopathy: A Case Report with Two Year Follow-up.
- [Background] Takla MK. Alterations of static and dynamic balance in patients with lumbar radiculopathy. Bulletin of Faculty of Physical Therapy. 2019;24:49-55.
- [Background] Kim KH, Leem MJ, Yi TI, Kim JS, Yoon SY. Balance Ability in Low Back Pain Patients With Lumbosacral Radiculopathy Evaluated With Tetrax: A Matched Case-Control Study. Ann Rehabil Med. 2020 Jun;44(3):195-202. doi: 10.5535/arm.19101. Epub 2020 May 29. PMID 32475097
- [Background] Das S, Dowle P, Iyengar R. Effect of spinal mobilization with leg movement as an adjunct to neural mobilization and conventional therapy in patients with lumbar radiculopathy: Randomized controlled trial. J Med Sci Res. 2018;6(1):11-9.
- [Background] Bello B, Danazumi MS, Kaka B. Comparative Effectiveness of 2 Manual Therapy Techniques in the Management of Lumbar Radiculopathy: A Randomized Clinical Trial. J Chiropr Med. 2019 Dec;18(4):253-260. doi: 10.1016/j.jcm.2019.10.006. Epub 2020 Sep 3. PMID 32952470
- [Background] Berry JA, Elia C, Saini HS, Miulli DE. A Review of Lumbar Radiculopathy, Diagnosis, and Treatment. Cureus. 2019 Oct 17;11(10):e5934. doi: 10.7759/cureus.5934. PMID 31788391
- [Background] Deng A, Wei L, Espiridion E. Assessing Nerve Block and Opioid Analgesics on Anxiety and Depression in Patients with Lumbar Radiculopathy. 2025.